CLINICAL TRIAL: NCT00087594
Title: An Open-Label, Multi-Center, Randomized, Safety, Feasibility and Tolerability Pilot Study of Pegasys® (Peginterferon Alfa-2a) Plus Copegus® (Ribavirin) in Previous Intravenous Drug Users Who Are Currently Enrolled in a Methadone Maintenance Treatment Program.
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Combination With Copegus (Ribavirin) in Patients With Chronic Hepatitis C (CHC) Enrolled in a Methadone Maintenance Treatment Program.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17251
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- Direct Observed Therapy (Experimental): Participants will receive the peginterferon alfa-2a plus ribavirin at the clinic as: subcutaneous peginterferon alfa-2a 180 microgram (mcg) (once in a week) for 24 weeks for Genotype 2 or 3 (G2/3), and for 48 weeks for Genotype 1 (G1); oral ribavirin 800 milligram (mg)/day (twice in a day) for 24 weeks for G2/3, and 1000 or 1200 mg/day (twice in a day) for 48 weeks for G1.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin
- Self-Administration Therapy (Experimental): Participants will receive the peginterferon alfa-2a plus ribavirin at home as: subcutaneous peginterferon alfa-2a 180 mcg (once in a week) for 24 weeks for G2/3, and for 48 weeks for G1; oral ribavirin 800 mg/day (twice in a day) for 24 weeks for G2/3, and 1000 or 1200 mg/day (twice in a day) for 48 weeks for G1.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 24 weeks (G 2/3) or 48 weeks (G 1)
Drug: ribavirin — 1000/1200mg (< or >= 75 kg, respectively), po in two doses daily for 48 weeks (G 1) or 800 mg po in two doses daily for 24 weeks (G 2/3)

SUMMARY:
This study will evaluate the safety and tolerability of PEGASYS plus ribavirin in previous intravenous (iv) drug users who have CHC and are currently enrolled in a methadone maintenance treatment program. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age
* CHC infection, genotype 1, 2, or 3
* naive to treatment for CHC infection
* enrolled in a methadone maintenance program with documented attendance for at least 3 months
* use of 2 forms of contraception during the study on both men and women

Exclusion Criteria:

* previous treatment for CHC infection
* co-infection with human immunodeficiency virus (HIV)
* current use of IV or other illicit drugs
* decompensated cirrhosis
* women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (7):
  - San Francisco, California
  - Farmington, Connecticut
  - Honolulu, Hawaii
  - Downers Grove, Illinois
  - Baltimore, Maryland
  - New York, New York
  - Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants were screened at 6 study sites in the United States (U.S) between 20 November 2003 and 25 September 2006.
Groups:
- Direct Observed Therapy: Participants received the peginterferon alfa-2a plus ribavirin at the clinic as: subcutaneous peginterferon alfa-2a 180 microgram (mcg) (once in a week) for 24 weeks for Genotype 2 or 3 (G2/3), and for 48 weeks for Genotype 1 (G1); oral ribavirin 800 milligram (mg)/day (twice in a day) for 24 weeks for G2/3, and 1000 or 1200 mg/day (twice in a day) for 48 weeks for G1.
- Self-Administration Therapy: Participants received the peginterferon alfa-2a plus ribavirin at home as: subcutaneous peginterferon alfa-2a 180 mcg (once in a week) for 24 weeks for G2/3, and for 48 weeks for G1; oral ribavirin 800 mg/day (twice in a day) for 24 weeks for G2/3, and 1000 or 1200 mg/day (twice in a day) for 48 weeks for G1.
Period: Overall Study
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Started | 24 | 24
Completed | 16 | 12
Not Completed | 8 | 12
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lack of Efficacy | 2 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all enrolled participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Observed Therapy | Self-Administration Therapy | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (10.50) | 46.8 (9.45) | 47.4 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Completion Rate (TCR)
Description: TCR is defined as the number of participants who completed the prescribed duration of the study treatment. TCR for G1 participants is defined as the number of participants who had a missing value or >= 2-log10 decrease in Hepatitis C virus-ribonucleic acid (HCV RNA) at Week 12 and completed 48 weeks of study treatment or had a < 2-log10 decrease from baseline at Week 12 and completed at least 12 weeks of study treatment. TCR for G2/ 3 participants is defined as the number of participants who completed 24 weeks of study treatment.
Time Frame: Up to 24 weeks for G2/3; up to 48 weeks for G1
Population: Safety Population included all participants who received at least one dose of study treatment and have at least one post-baseline safety assessment (adverse event, laboratory/vital sign, physical examination; Beck Depression Inventory; Hepatitis Quality-of-Life Questionnaire). n = number of participants at indicated time points for each arm.
Measure: Number; unit: participants
Groups:
- Direct Observed Therapy: Participants received the peginterferon alfa-2a plus ribavirin at the clinic as: subcutaneous peginterferon alfa-2a 180 mcg (once in a week) for 24 weeks for Genotype 2 or 3 (G2/3), and for 48 weeks for Genotype 1 (G1); oral ribavirin 800 mg/day (twice in a day) for 24 weeks for G2/3, and 1000 or 1200 mg/day (twice in a day) for 48 weeks for G1.
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  G1 (n = 13, 16) | 9 | 10
  G1, 2 log drop at Week 12 (n = 4, 9) | 4 | 5
  G1, non 2 log drop at Week 12 (n = 4, 4) | 4 | 4
  G1, missing HCV-RNA at Week 12 (n = 5, 3) | 1 | 1
  G2/3 (n = 11, 8) | 11 | 7
Statistical Analysis 1: Comparison: Direct Observed Therapy vs Self-Administration Therapy; 95% CI for G1 participants; Test type: Superiority or Other; Difference = 7, 95% CI 2-sided [-27.8 to 41.3]
Statistical Analysis 2: Comparison: Direct Observed Therapy vs Self-Administration Therapy; 95% CI for G2/3 participants; Test type: Superiority or Other; Difference = 13, 95% CI 2-sided [-10.4 to 35.4]
Statistical Analysis 3: Comparison: Direct Observed Therapy vs Self-Administration Therapy; 95% CI for G1 participants with 2 log drop at W 12; Test type: Superiority or Other; Difference = 44, 95% CI 2-sided [12.0 to 76.9]
Statistical Analysis 4: Comparison: Direct Observed Therapy vs Self-Administration Therapy; 95% CI for G1 participants with non 2 log drop at W 12; Test type: Superiority or Other; Difference = 0
Statistical Analysis 5: Comparison: Direct Observed Therapy vs Self-Administration Therapy; 95% CI for G1 participants with missing HCV-RNA at W 12; Test type: Superiority or Other; Difference = -13, 95% CI 2-sided [-77.2 to 50.5]

2. Secondary Outcome: Number of Participants With Sustained Virological Response (SVR) Rate at 24 Weeks Post Treatment (Week 48 for G2/3 and Week 72 for G1)
Description: SVR is defined as the number of participants with undetectable HCV-RNA (< 10 international unit per milliliter [IU/mL]) at 24 weeks post treatment completion.
Time Frame: Week 48 for G2/3 and Week 72 for G1
Population: ITT Population included all enrolled participants who received at least one dose of study medication. n = number of participants at indicated time points for each arm.
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  G1 (n = 13, 16) | 4 | 5
  G2/3 (n = 11, 8) | 10 | 2

3. Secondary Outcome: Number of Participants With Virological Response Rate at Weeks 12, 24, and 48 (G1 Only) During Treatment and at 12 Weeks After Treatment Completion
Description: Virological Response Rate is defined as the number of participants with undetectable HCV-RNA (< 10 IU/mL). Treatment completion (end of treatment [EOT]) for G1 was Week 48 and for G2 or 3 was Week 24.
Time Frame: Weeks 12, 24, and 48 for G1 and Weeks 12 and 24 for G2/3; 12 and 24 weeks after EOT for G1 (Weeks 60 and 72) and G2/3 (Weeks 36 and 48)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Week 12 (G1), (n = 13, 16) | 3 | 5
  Week 24 (G1), (n = 13, 16) | 5 | 8
  Week 48 (EOT) (G1), (n = 13, 16) | 5 | 8
  12 weeks after EOT (G1), (n = 13, 16) | 5 | 4
  Week 12 (G2/3), (n = 11, 8) | 11 | 8
  Week 24 (EOT) (G2/3), (n = 11, 8) | 11 | 7
  12 Weeks after EOT (G2/3), (n = 11, 8) | 9 | 3

4. Secondary Outcome: Number of Participants With Biochemical Response Rate at Weeks 12, 24, and 48 (G1 Only) During Treatment and at 12 and 24 Weeks After Treatment Completion
Description: Biochemical response is defined as the number of participants with a normal serum alanine aminotransferase (ALT) concentration (i.e., ALT < 30 U/L). EOT for G1 was Week 48 and for G2/3 was Week 24.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Week 12 (G1), (n = 13, 16) | 3 | 13
  Week 24 (G1), (n = 13, 16) | 5 | 13
  Week 48/EOT (G1), (n = 13, 16) | 4 | 5
  12 Weeks after EOT (G1), (n = 13, 16) | 6 | 8
  24 Weeks after EOT (G1), (n = 13, 16) | 4 | 7
  Week 12 (G2/3), (n = 11, 8) | 10 | 2
  Week 24/EOT (G2/3), (n = 11, 8) | 10 | 4
  12 Weeks after EOT (G2/3), (n = 11, 8) | 10 | 4
  24 Weeks after EOT (G2/3), (n = 11, 8) | 11 | 3

5. Secondary Outcome: Number of Participants With > =2 Log Drop From Baseline or Undetectable HCV-RNA (<10 IU/mL) at Week 12
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Week 12 (G1), (n = 13, 16) | 4 | 9
  Week 12 (G2/3), (n = 11, 8) | 11 | 8

6. Secondary Outcome: Mean Absolute Score of Beck Depression Inventory, Second Edition (BDI-II)
Description: BDI-II is 21-item self-report instrument to assess severity of symptoms of depression. There is a four-point scale for each item ranging from 0 to 3. Degrees of depression defined by the total BDI-II score as: minimal (0 to 13), mild (14 to 19), moderate (20 to 28), and severe depression (>= 29). Higher scores reflective of greater severity (worse outcome).
Time Frame: Baseline (Day -30 to -1), EOT visit (Week 24 for G2/3 and Week 48 for G1), and end of study (EOS) visit (Week 48 for G2/3 and Week 72 for G1).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline, (n = 24, 24) | 8.7 (1.2) | 8.6 (0.9)
  EOT (Week 24/48), (n = 18, 13) | 13.6 (2.4) | 22.8 (3.0)
  EOS (Week 48/72), (n = 22, 19) | 8.6 (2.0) | 13.4 (2.4)

7. Secondary Outcome: Mean Change From Baseline in BDI-II Score to EOT (Week 24/48) and EOS (Week 48/72) Visits
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
units on a scale
  EOT (Week 24/48), (n = 18, 13) | 6.1 (2.2) | 13.5 (3.2)
  EOS (Week 48/72), (n = 22, 19) | 0.4 (1.8) | 4.5 (2.4)

8. Secondary Outcome: Number of Participants With Degrees of Depression as Defined by the BDI-II Score
Description: Participants with degrees of depression as defined by the BDI-II Score were reported. BDI-II is 21-item self-report instrument to assess severity of symptoms of depression. There is a four-point scale for each item ranging from 0 to 3. Degrees of depression defined by the total BDI-II score as: minimal (0 to 13), mild (14 to 19), moderate (20 to 28), and severe depression (>= 29). Higher scores reflective of greater severity (worse outcome).
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Baseline, none-mild | 22 | 24
  Baseline, moderate | 2 | 0
  Highest post-baseline, none-mild | 16 | 9
  Highest post-baseline, moderate | 5 | 11
  Highest post-baseline, severe | 3 | 3
  Last post-baseline, none-mild | 20 | 18
  Last post-baseline, moderate | 3 | 3
  Last post-baseline, severe | 1 | 2

9. Secondary Outcome: Mean Absolute Scores for Hepatitis Quality-of-Life Questionnaire (HQLQ) at EOT (Week 24/48) Visit and 24 Weeks After EOT Visit
Description: The HQLQ is a multiple-choice questionnaire includes the eight individual qualify-of-life scales of the Medical Outcomes Study 36-item Short-form Health Survey as: Social functioning (SF), role limitations due to emotional problems (RE), vitality (VT), general mental health (MH), physical functioning (PF), role limitations due to physical problems (RP), freedom from bodily pain (BP), and general health (GH). In addition, two other generic scales (positive well-being [PWB] and health distress [HD]) and two hepatitis-specific scales (limitations because of chronic hepatitis C [HLIM] and health distress because of chronic hepatitis C [HHD]) were included. Scores were scaled to a 0 to 100 range, with 0 = bad and 100 = good. A higher score indicates an improvement.
Time Frame: Baseline (Day -30 to -1), 24 weeks after EOT visit (Week 48 for G2/3 and Week 72 for G1)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
units on a scale
  SF at Baseline (n = 23, 24) | 70.7 (4.1) | 75.5 (5.2)
  SF at EOT, (n = 15, 12) | 50.0 (7.0) | 35.4 (8.9)
  SF at 24 Weeks after EOT, (n = 17, 15) | 72.8 (6.8) | 59.2 (8.4)
  RE at Baseline (n = 23, 24) | 55.1 (9.0) | 75.0 (7.0)
  RE at EOT, (n = 14, 12) | 47.6 (12.0) | 36.1 (12.6)
  RE at 24 Weeks after EOT, (n = 17, 15) | 74.5 (9.7) | 62.2 (11.7)
  MH at Baseline (n = 23, 24) | 63.7 (3.4) | 73.5 (3.6)
  MH at EOT, (n = 15, 12) | 53.6 (5.9) | 51.7 (5.6)
  MH at 24 Weeks after EOT, (n = 17, 15) | 67.5 (6.1) | 57.9 (4.7)
  PF at Baseline (n = 23, 24) | 74.6 (4.9) | 80.0 (4.6)
  PF at EOT, (n = 15, 12) | 59.0 (8.4) | 52.9 (8.3)
  PF at 24 Weeks after EOT, (n = 17, 14) | 75.9 (6.0) | 62.9 (8.8)
  RP at Baseline (n = 23, 24) | 62.0 (8.1) | 59.4 (8.8)
  RP at EOT, (n = 15, 12) | 26.7 (9.6) | 16.7 (7.1)
  RP at 24 Weeks after EOT, (n = 17, 14) | 66.2 (9.3) | 55.4 (11.5)
  BP at Baseline (n = 23, 24) | 67.0 (4.6) | 72.2 (4.1)
  BP at EOT, (n = 14, 12) | 55.9 (5.6) | 47.8 (6.9)
  BP at 24 Weeks after EOT, (n = 17, 15) | 66.7 (6.0) | 68.1 (7.3)
  GH at Baseline (n = 23, 24) | 56.3 (2.8) | 60.8 (4.0)
  GH at EOT, (n = 15, 12) | 54.0 (5.3) | 37.2 (4.4)
  GH at 24 Weeks after EOT, (n = 17, 15) | 58.7 (6.5) | 46.6 (5.4)
  VT at Baseline (n = 23, 24) | 48.0 (4.2) | 52.7 (3.8)
  VT at EOT, (n = 15, 12) | 29.0 (4.6) | 20.0 (4.8)
  VT at 24 Weeks after EOT, (n = 17, 15) | 54.4 (6.9) | 41.3 (5.9)
  HD at Baseline (n = 23, 24) | 65.7 (4.9) | 76.9 (4.5)
  HD at EOT, (n = 15, 12) | 62.3 (5.7) | 43.3 (7.8)
  HD at 24 Weeks after EOT, (n = 17, 15) | 73.8 (6.8) | 52.7 (7.3)
  PWB at Baseline (n = 23, 24) | 50.0 (4.4) | 40.2 (4.3)
  PWB at EOT, (n = 15, 12) | 65.3 (5.5) | 63.8 (5.6)
  PWB at 24 Weeks after EOT, (n = 17, 15) | 45.3 (6.7) | 47.0 (6.6)
  HLIM at Baseline (n = 23, 23) | 74.5 (6.0) | 76.8 (6.1)
  HLIM at EOT, (n = 15, 12) | 59.1 (7.4) | 40.0 (8.7)
  HLIM at 24 Weeks after EOT, (n = 16, 15) | 84.2 (5.6) | 68.9 (9.6)
  HHD at Baseline (n = 23, 23) | 62.8 (5.5) | 69.8 (5.7)
  HHD at EOT, (n = 15, 12) | 58.7 (8.2) | 50.4 (7.4)
  HHD at 24 Weeks after EOT, (n = 16, 15) | 81.6 (6.0) | 67.3 (7.3)

10. Secondary Outcome: Number of Participants With Compliance to the Prescribed Treatment Regimen
Description: Participants with compliance to the prescribed treatment regimen for peginterferon alfa-2a and ribavirin was reported. Compliance was calculated as (total cumulative dose taken) / (total cumulative original dose prescribed for the entire study) x 100. Total treatment duration = Maximum doses of peginterferon alfa-2a and ribavirin in days / (48*7) for G1, total treatment duration = Maximum doses of peginterferon alfa-2a and ribavirin in days / (24*7) for G2/3.
Time Frame: Up to Week 24 for G 2/3; up to Week 48 for G1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Peginterferon alfa-2a, 0-60% | 8 | 8
  Peginterferon alfa-2a, >60-80% | 0 | 1
  Peginterferon alfa-2a, >80-97% | 1 | 4
  Peginterferon alfa-2a, >97% | 15 | 11
  Ribavirin, 0-60% | 8 | 10
  Ribavirin, >60-80% | 4 | 1
  Ribavirin, >80-97% | 5 | 7
  Ribavirin, >97% | 7 | 6
  Total Treatment Duration, 0-60% | 8 | 8
  Total Treatment Duration, >60-80% | 0 | 1
  Total Treatment Duration, >80-97% | 1 | 3
  Total Treatment Duration, >97% | 15 | 12

11. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital Signs included systolic blood pressures (SBP), diastolic blood pressures (DBP), and pulse rate (PR). Abnormal vital signs were reported as low or high abnormal. It was defined as < 85 mm Hg or > 180 mm Hg with a change from baseline of > 20%; DBP as > 110 mm Hg with a change from baseline of > 20%; and PR as < 50 bpm and > 120 bpm with a change from baseline of > 20%.
Time Frame: Up to 24 weeks of treatment-free follow-up visit (Week 48 for G2/3 and Week 72 for G1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  SBP - High | 1 | 0
  SBP - Low | 1 | 0
  DBP - High | 2 | 0
  PR - Low | 1 | 1

12. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities (Hematology)
Description: Hematology included hematocrit (fraction), hemoglobin, platelets count, Red blood cells (RBC), White blood cell (WBC), eosinophils, lymphocytes, monocytes, neutrophils, Partial Thromboplastin time (PTT), Prothrombin Time International Normalized Ratio (PT INR). Laboratory values falling outside the marked reference range as defined by Roche's "International Guideline for the Handling and Reporting of Laboratory Data", and were clinically relevant change from baseline were considered marked laboratory abnormalities. It was reported as low or high abnormal.
Time Frame: Up to 24 weeks post treatment (Week 48 for G2/3 and Week 72 for G1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Hematocrit (fraction) - Low (n = 24, 24) | 10 | 11
  Hemoglobin - Low (n = 24, 24) | 10 | 16
  Platelets - Low (n = 24, 24) | 11 | 10
  RBC - Low (n = 24, 24) | 14 | 18
  WBC - High (n = 24, 24) | 0 | 1
  WBC - Low (n = 24, 24) | 18 | 19
  Eosinophils - High (n = 24, 24) | 0 | 1
  Lymphocytes - Low (n = 24, 24) | 8 | 10
  Monocytes - High (n = 24, 24) | 0 | 1
  Neutrophils - High (n = 24, 24) | 0 | 4
  Neutrophils - Low (n = 24, 24) | 19 | 20
  PTT - High (n = 22, 23) | 2 | 3
  PT INR (ratio) - High (n = 22, 23) | 0 | 2

13. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities (Biochemistry)
Description: Laboratory values falling outside the marked reference range as defined by Roche's "International Guideline for the Handling and Reporting of Laboratory Data", and were clinically relevant change from baseline were considered marked laboratory abnormalities. It was reported as low or high abnormal.
Time Frame: Up to 24 weeks post treatment (Week 48 for G2/3 and Week 72 for G1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Aspartate aminotransferase - High (n = 24, 24) | 2 | 8
  Alanine aminotransferase - High (n = 24, 24) | 2 | 4
  Albumin - Low (n = 24, 24) | 0 | 4
  Total protein - High (n = 24, 24) | 1 | 1
  Total protein - Low (n = 24, 24) | 0 | 1
  Chloride - Low (n = 24, 24) | 2 | 3
  Sodium - Low (n = 24, 24) | 3 | 2
  Calcium - Low (n = 24, 24) | 0 | 5
  Phosphate - High (n = 24, 24) | 1 | 2
  Phosphate - Low (n = 24, 24) | 6 | 7
  Glucose random - High (n = 24, 24) | 1 | 2
  Triglycerides - High (n = 24, 24) | 9 | 6
  Thyroxine (T4) - High (n = 22, 22) | 4 | 2
  Thyroid-Stimulating Hormone - High (n = 22, 22) | 0 | 3

14. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), Any Serious Adverse Events (SAEs), and Study Discontinuation
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. Reason for discontinuation was categorized as safety and non-safety, where safety reasons included abnormality of laboratory tests, AEs, and death; and non-safety reasons included insufficient therapeutic response, early improvement, violation of selection criteria at entry, other protocol violation, refused treatment, failure to return and other. Participants who discontinued the study with any reason were recorded.
Time Frame: Up to 24 weeks post treatment (Week 48 for G2/3 and Week 72 for G1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Number analyzed (Participants) | 24 | 24
participants
  Any AEs | 24 | 24
  Any SAEs | 3 | 3
  AEs | 2 | 3
  Study discontinuation due to Insufficient Response | 2 | 5
  Study discontinuation due to Refused Treatment | 4 | 2
  Study discontinuation due to Failure to Return | 0 | 2

ADVERSE EVENTS:
Time Frame: From baseline to Week 72
Arm/Group | Direct Observed Therapy | Self-Administration Therapy
Serious Adverse Events (participants affected / at risk) | 3/24 | 3/24
Other Adverse Events (participants affected / at risk) | 24/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Direct Observed Therapy (N=24) | Self-Administration Therapy (N=24)
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Direct Observed Therapy (N=24) | Self-Administration Therapy (N=24)
Fatigue (General disorders) | 16 | 19
Irritability (General disorders) | 8 | 9
Chills (General disorders) | 6 | 7
Pyrexia (General disorders) | 5 | 8
Injection site erythema (General disorders) | 4 | 2
Asthenia (General disorders) | 3 | 2
Influenza like illness (General disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 13 | 14
Vomiting (Gastrointestinal disorders) | 6 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Depression (Psychiatric disorders) | 9 | 10
Insomnia (Psychiatric disorders) | 8 | 10
Anxiety (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 9 | 10
Dysgeusia (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 2
Mental impairment (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 8
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Tooth extraction (Surgical and medical procedures) | 0 | 2
Blood pressure increased (Investigations) | 2 | 0
Drug screen positive (Investigations) | 7 | 4
Haemoglobin decreased (Investigations) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.